CLINICAL TRIAL: NCT03890237
Title: Gender Transformative Programming to Improve Capabilities of Young Adolescents in Ethiopia: A Cluster Randomized Control Trial
Brief Title: GAGE Act With Her-Ethiopia Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Overseas Development Institute (Unknown); Addis Ababa University (Other); University of Oklahoma (Other); Pathfinder International (Industry); Care International (Unknown); UK Department for International Development on behalf of UK Aid (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Sarah Baird, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAGE AWH-E 2019
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Adolescent Behavior; Gender
MeSH Terms: conditions — Adolescent Behavior; Coitus | interventions — alpha 1-Antichymotrypsin

STUDY DESIGN:
Intervention Model Description: The impact evaluation study is a cluster-randomized controlled trial among 175 communities with five study arms: control (no intervention), AWH-E, Her Spaces, AWH- E + asset transfer, and AWH-E without community engagement and systems strengthening.
Masking Description: Study participants will not be masked to their assignment, but will not know the full set of treatment and comparison groups, or what those other groups receive. Given cluster level randomization, contamination will be minimized. Enumerators who collect the survey data that forms the basis of the evaluation will not be explicitly told the treatment status of a given Kebele, however, given the community level nature of the intervention it may be possible for them to ascertain whether it is a treatment or control Kebele. Statistical analyses will be done by the investigators who will not be masked to the treatment status of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Business as usual, no intervention
- Her Spaces (Experimental): Starts in year 1; intervention package with 11-13 year old girls for 10 months; standard parental and community engagement. All programming ends after 10 months.
  Interventions: Behavioral: Her Spaces
- Act With Her (Experimental): Starts in year 1; core intervention package with 10-13 year old girls and boys for 10 months; 6 dedicated sessions with parents; and community-level system strengthening up to 24 months.
  Interventions: Behavioral: Act With Her
- Act With Her + Asset Transfer (Experimental): Starts in year 1; core intervention package with 10-13 year old girls and boys for 10 months; asset transfer for girls over 10 months; 6 dedicated sessions with parents; and community-level system strengthening up to 24 months.
  Interventions: Behavioral: Act With Her + Asset Transfer
- Act With Her (simple) (Experimental): Starts in year 1; core intervention package with 10-13 year old girls and boys for 10 months; 6 dedicated sessions with parents; does not include community-level systems strengthening. All programming ends after 10 months.
  Interventions: Behavioral: Act With Her (simple)

INTERVENTIONS:
Behavioral: Her Spaces — Her Spaces will comprise a set of activities leveraging the Her Spaces curriculum and program model which includes curriculum-based sessions for 11-13 year old girls, with 40 sessions delivered weekly over the course of 10 months
  Arms: Her Spaces
Behavioral: Act With Her — Act With Her was designed to facilitate adolescent transitions to adulthood via improvements across the six GAGE domains (education, bodily integrity, health, psychosocial well-being, voice and agency, and economic empowerment). Project activities fall into three main categories: curriculum-based programming with adolescent girls and boys, community transformation, and systems strengthening. Act With Her will work with 10-13 year old girls and boys for 10 months and implement community-level and high-level system strengthening work up to 24 months (in rural and pastoralist areas).
  Arms: Act With Her
Behavioral: Act With Her + Asset Transfer — This arm will implement the Act With Her program described above, using program curricula with 10-13-year-old girls and boys over 10 months and conducting community-level systems strengthening up to 24 months. Additionally, the girls participating in this arm will receive one of three asset transfer options. The packages will be of equal value (115 USD) - one will include school supplies, one will include hygiene supplies, and will be a combination of both. Each adolescent girl will choose which package she would like to receive and will receive components of the package at 3 timepoints over the course of the first 10 months of the project.
  Arms: Act With Her + Asset Transfer
Behavioral: Act With Her (simple) — This arm will implement the Act With Her curricula described above with 10-13 year old girls and boys over 10 months. The adolescent groups will follow the same model (near-peer, same-sex mentors, 40 weekly meetings for girls, 18 meetings for boys, 4 of which are joint sessions for boys and girls, 6 sessions for parents), but will not include community-level systems strengthening activities
  Arms: Act With Her (simple)

SUMMARY:
This study evaluates the impact of Act With Her Ethiopia (AWH-E), a gender transformative multi-level program that aims to improve the lives of young adolescent boys and girls.

DETAILED DESCRIPTION:
Unequal gender norms and power dynamics are often driven and reinforced by adolescent girls' male peers, families, communities, and the broader institutional structures that surround them. Without change in gender attitudes and norms at each of these levels, improved outcomes for key transitions are much less likely to be sustained. Efforts to nurture change must also acknowledge that adolescents' opportunities and capabilities are shaped by complex, intersectional forces including ethnicity, caste, religion, and disability, among others. This multi-arm randomized control trial aims to improve the evidence base on effective approaches to improve multi-sectoral outcomes for girls across the following domains from the Gender and Adolescence: Global Evidence (GAGE) framework: education and learning; health, nutrition and sexual and reproductive health; bodily integrity; psychosocial well-being; voice and agency; and economic empowerment.

Specifically, the trial has four goals:

1. To evaluate the impact of Act With Her in Ethiopia (AWH-E) - a gender-transformative multi-level program - on young adolescent girls' and boys' capabilities (11-13) in the short- and long-run across the six GAGE capability domains using a multi-arm cluster randomized control trial across two regions (Amhara and Oromia).
2. To compare the impact of AWH-E to a more basic gender-synchronized program (AWH-E without community engagement and systems strengthening), a standalone girls' group program (Her Spaces), and the gender-transformative program with economic support (AWH-E + Asset Transfers) on young adolescent capability achievements and transitions in the short- and longer- terms across two regions (Amhara and Oromia).
3. To evaluate the impact of AWH-E on young adolescent capability achievements and transitions in the short- and long- term in pastoralist contexts (Afar).
4. To use mixed-methods research to understand the mechanisms driving the impact, and in particular what works, for whom, and why.

ELIGIBILITY:
Inclusion Criteria:

* girls and boys 10-13 at time of enrollment in Act With Her Arms
* girls 11-13 female at time of enrollment in Her Spaces Arm

Exclusion Criteria:

* None

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Both males and females are eligible for the program, but the specific programming is different for males and females. In Her Spaces arms there is no male specific programming.
Enrollment: 4500 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Standardized Index of Education and Learning (girls) | 20 months after intervention starts
  Standardized index of education and learning at the individual level. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. The index is comprised of four components: indicator for enrolled in school (at time in survey, or if school not in session at survey, at time of most recent session), share of school days attended (past two weeks; among those enrolled), indicator for did not miss more than one week of school at one time (past 12 months; among those enrolled), aspires for secondary degree or higher. The construction of the index, and a detailed description of its components is described in the protocol.
Standardized index of Bodily Integrity (girls) | 20 months after the intervention starts
  Standardized index of bodily integrity at the individual level. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. The index is comprised of six indicators: peer violence scale (past 12 months, inverse), indicator for did not experience peer violence (past 12 months), indicator for did not perpetrate peer violence (past 12 months), indicator for did not experience violence or witness violence against female caregiver in the household (past 12 months), indicator for did not experience sexual violence (past 12 months), ideal age of marriage. The construction of the index, and a detailed description of its components is described in the protocol.
Standardized Index of Health, Nutrition, and Sexual and Reproductive Health (girls) | 20 months after the intervention starts
  Standardized index of bodily integrity at the individual level. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. The index is comprised of five components: indicator for self-reported health very good or good, proportion of meals yesterday with meat/chicken/fish/egg, indicator if ever hungry because not enough food (past four weeks), indicator for normal activities not affected during menstruation (among those who have reached menarche), index of improved menstrual hygiene practices (among those who have reached menarche), ideal age of first child (among childless). The construction of the index, and a detailed description of its components is described in the protocol.
Standardized Index of Psychosocial Well-Being (girls) | 20 months after the intervention starts
  Standardized index of bodily integrity at the individual level. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. The index is composed of three components. Rosenberg Self Esteem Scale score, General Health Questionnaire-12 (GHQ-12; measure of psychosocial distress; inverse) score, Child and Youth Resilience Scale score. The construction of the index, and a detailed description of its components is described in the protocol
Standardized Index of Voice and Agency (girls) | 20 months after the intervention starts
  Standardized index of voice and agency. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. The index is composed of five components: index of participation in decision making (school, family; standardized separately for in school and out of school), index of comfort discussing issues, index of voice, index of mobility, index of collective action. The construction of the index, and a detailed description of its components is described in the protocol.
Standardized Index of Economic Empowerment (girls) | 20 months after the intervention starts
  Standardized index of economic empowerment. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. Index is comprised of five components: indicator for any control of money (past 12 months), indicator for any savings for the future, indicator for aspires to be employed in skilled or professional work when adult, aspires to have employment or a business when adult, proportion of time yesterday in leisure and school (including travel to and from, and studying). The construction of the index, and a detailed description of its components is described in the protocol.
Standardized Index of Cross-Cutting Gender Issues (girls) | 20 months after the intervention ends
  Standardized index of cross-cutting gender issues. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. Index is comprised of six components: index of gender equitable attitudes, index of gender consciousness, index of trusted friends (supportive social network), indicator for supportive adult, knowledge index, index of access to health services. The construction of the index, and a detailed description of its components is described in the protocol.
Standardized Index of Cross-Cutting Gender Issues (boys) | 20 months after the intervention ends
  Standardized index of cross-cutting issues for boys. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. Index of composed of 9 components: index of gender equitable attitudes, index of gender consciousness, index of gender equitable behaviors, indicator for not perpetrating peer violence, peer violence index (inverse), indicator for not being a victim of peer violence, General Health Questionare-12 (GHQ-12; measure of mental health, inverse) score, indicator for supportive adult, knowledge index. The construction of the index, and a detailed description of its components is described in the protocol
Standardized Index of Cross-cutting Gender Issues (primary female caregivers of girls) | 20 months after the intervention ends
  Standardized index of cross-cutting issues for primary female caregivers of girls. The index is standardized to be mean 0 standard deviation 1. Higher values are better outcomes. Each component of the index is also standardized to be mean zero standard deviation one before summing. Index consists of 8 components: aspiration for adolescent's education, expected age of marriage for adolescent, aspiration for adolescent to work in skilled or professional employment as an adult, aspiration for adolescent to be employed or own a business as an adult, index of support for education, indicator for did not cut back food same for boys and girls (past 4 weeks), index of gender consciousness, index of gender attitudes. The construction of the index, and a detailed description of its components is described in the protocol

CONTACTS AND LOCATIONS:
Locations (3):
- Ethiopia (3):
  - Zone 5, Afar Region
  - South Gondar, Amhara
  - East Hararghe, Oromiya

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be made public through the UK data archive per DfID funding requirements.